CLINICAL TRIAL: NCT01185444
Title: Efficacy of 3 Weekly Injections of a Bacterial-- Sourced Hyaluronate on Pain and Physical Function in Patients With Knee Osteoarthritis-a Randomized Controlled Clinical Trial
Brief Title: Efficacy of Three Weekly Injections of a Bacterial-- Sourced Hyaluronate on Pain and Function in Patients With Knee Osteoarthritis (OA)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Kaohsiung Veterans General Hospital. (Other)
Responsible Party: Kaohsiung Veterans General Hospital, Kaohsiung Veterans General Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: VGHKS97-CT9-12
Record Dates: First submitted 2010-08-13; First posted 2010-08-20 (Estimated); Last update posted 2010-08-20 (Estimated); Status verified 2008-12

CONDITIONS: Hyaluronate; Osteoarthritis; Knee
Keywords: Knee Balance; Hyaluronate; Osteoarthritis; Viscosupplementation
MeSH Terms: conditions — Osteoarthritis | interventions — Hyaluronic Acid

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Hya-Joint (Experimental): The Hya-Joint group received 3 weekly intraarticular injections of 2 ml sodium hyaluronate (Hya-Joint, derived from Streptococcus zooepidemicus and produced by a highly purified biologic fermentation process, molecular weight 650-1200 kDa),into the target knee.
  Interventions: Procedure: Hya-Joint
- Hyalgan (Active Comparator): the control group received 3 weekly intraarticular injections of 2 ml sodium hyaluronate (, extracted from chicken combs, molecular weight 500-730kDa) into the knee joints.
  Interventions: Procedure: Hyalgan

INTERVENTIONS:
Procedure: Hya-Joint — The Hya-Joint group received 3 weekly intraarticular injections of 2 ml sodium hyaluronate (Hya-Joint, derived from Streptococcus zooepidemicus and produced by a highly purified biologic fermentation process, molecular weight 650-1200 kDa),into the target knee.
  Arms: Hya-Joint
Procedure: Hyalgan — The control group received 3 weekly intraarticular injections of 2 ml sodium hyaluronate (Hyalgan, extracted from chicken combs, molecular weight 500-730kDa) into the knee joints.
  Arms: Hyalgan

SUMMARY:
Three weekly injections of hyaluronate (Hya-Joint) are safe and well tolerated, provide rapid pain relief as early as 1 and 2 weeks after the first injection, and improve function in patients with knee osteoarthritis. The treatment effects can last for 6 months.

DETAILED DESCRIPTION:
Background: Viscosupplementation with intra-articular hyaluronate injections is a safe and effective treatment of knee osteoarthritis. There are several forms of hyaluronate with different origin, method of production, molecular weight, dosing instructions and possibly clinical outcomes. Most current hyaluronate products are avian in origin, and only few are bioengineered via bacterial fermentation. The purpose of this study was to evaluate the efficacy and safety of 3 weekly injections of a bacterial-sourced hyaluronate (Hya-Joint) in patients with knee osteoarthritis.

Methods: As a prospective randomized observer-blind study done in a university-affiliated tertiary care medical center, patients with knee osteoarthritis for at least 6 months were enrolled. Eligible patients were randomized to receive three weekly intraarticular injections of either bacterial-sourced hyaluronate (Hya-Joint) or avian-derived hyaluronate (Hyalgan) into the target knee. The primary outcome was the visual analog scale (VAS) change from baseline for knee pain at 6-month follow-up. Secondary outcome measures included Lequesne index, timed up and go test (TUG), patients' global satisfaction and analgesics consumption.

Results: A total of 95 participants were randomly assigned and 89 participants completed the study. Both groups had significant improvements in pain as early as 1 and 2 weeks after the first injection, and the pain-reduction effects could last for 6 months, with no between-group differences. The Lequesne index scores and results of TUG tests improved significantly from baseline in both group at all follow-up visits (p<0.001 for each test compared with baseline), with no significant between-group differences at 1-month and 6-month follow-up. However, significantly greater improvements favoring the Hya-Joint group were noted at 3-month follow-up (p<0.05). No between-group differences were seen regarding the use of analgesics. Both groups reported high satisfaction at 6-month follow-up. No serious adverse events occurred.

Conclusions: Three weekly injections of hyaluronate (Hya-Joint) are safe and well tolerated, provide rapid pain relief as early as 1 and 2 weeks after the first injection, and improve function in patients with knee osteoarthritis. The treatment effects can last for 6 months.

ELIGIBILITY:
Inclusion Criteria:

* (1) age 40 years or older, presence of a primary knee OA with knee pain for at least 6 months despite conservative treatment (rest, physical therapy, orthoses or pain medications etc.); (2) had average pain on knee movement of at least 3 cm on a 10-cm VAS; (3) had a current Lequesne index score (described below) >7 (possible range, 0-24); (4) were willing to discontinue all nonsteroidal anti-inflammatory drugs (NSAIDs) or other analgesic medication (except for rescue medication) for the duration of the study; and (5) were willing to not receive physical therapy or trial of shoe modifications or orthoses during the study period.

Exclusion Criteria:Exclusion criteria included previous orthopedic surgery on the spine or lower limbs, knee instability or marked deformity on examination, clinically apparent tense effusion of the knee, intra-articular steroid or HA injection in any joint within the past 6 months, and concomitant inflammatory arthropathy or other rheumatologic, neurological, cardiovascular or psychiatric disorders that would interfere with the clinical assessment during the study period.

-

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 89 (Actual)
Dates: Start 2009-02; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
visual analog scale | 6 months after the third injection
  The patient rated the intensity of pain with regard to average pain on knee movement over the previous week using a 10-cm horizontal VAS (10-cm line; 0= no pain to 10= worst imaginable pain)

SECONDARY OUTCOMES:
Lequesne index | 6 months after the third injection
  Lequesne index was used to assess severity of knee symptoms during the last week23. It is validated and includes the measurement of pain (5 items), walking distance (2 items), and activities of daily living (4 items). Maximal score is 24 and higher scores represent worse function
Timed " Up-and-Go" test | 6 months after the third injection.
  Timed " Up-and-Go" test (TUG) is a simple test of basic physical functional mobility for frail elderly persons with high interrater reliability and content reliability24. A patient is asked to rise from an armchair, walk 3 meters at a safe and comfortable pace, turn around, walk back to the chair, and sit down again. The whole procedure is demonstrated first before the actual test. The score is the time in seconds it takes to complete these tasks
the level of global satisfaction | 6 months after the third injection.
  Patients were asked to rate the level of global satisfaction compared to their preinjection condition at each follow-up visit. The rating was based on a 7-point categorical scale weighted from completely satisfied, satisfied, somewhat satisfied, no change, somewhat dissatisfied, dissatisfied to completely dissatisfied.

CONTACTS AND LOCATIONS:
Overall Officials: Shu-Fen Sun, MD, Principal Investigator — Veterans General Hospital, Kaohsiung;National Yang-Ming University School of Medicine, Taiwan; Chien-Wei Hsu, MD, Principal Investigator — Department of Internal Medicine, Kaohsiung Veterans General Hospital; Hsien-Pin Sun, MD, Principal Investigator — Cheng Ching Hospital, Taiwan; Hung-Ju Li, MS, Principal Investigator — Institute of Statistics, National University of Kaohsiung, Taiwan; Jue-Long Wang, MD, Principal Investigator — Kaohsiung Veterans General Hospital, Taiwan
Locations (1):
- Department of Physical Medicine and Rehabilitation, Veterans General Hospital,, Kaohsiung City, Taiwan

REFERENCES:
- [Background] Sun SF, Hsu CW, Hwang CW, Hsu PT, Wang JL, Tsai SL, Chou YJ, Hsu YW, Huang CM, Wang YL. Hyaluronate improves pain, physical function and balance in the geriatric osteoarthritic knee: a 6-month follow-up study using clinical tests. Osteoarthritis Cartilage. 2006 Jul;14(7):696-701. doi: 10.1016/j.joca.2006.01.010. Epub 2006 Mar 6. PMID 16520067
- [Background] Adams ME, Atkinson MH, Lussier AJ, Schulz JI, Siminovitch KA, Wade JP, Zummer M. The role of viscosupplementation with hylan G-F 20 (Synvisc) in the treatment of osteoarthritis of the knee: a Canadian multicenter trial comparing hylan G-F 20 alone, hylan G-F 20 with non-steroidal anti-inflammatory drugs (NSAIDs) and NSAIDs alone. Osteoarthritis Cartilage. 1995 Dec;3(4):213-25. doi: 10.1016/s1063-4584(05)80013-5. PMID 8689457